CLINICAL TRIAL: NCT04251650
Title: Search for a Microbiotic Signature Associated With Periodontitis According to the Chicago Classification 2018
Brief Title: PAROMIP Pilot Study PAROdontites & MIcrobiota Periodontal
Acronym: PAROMIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 30042019
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Periodontitis
Keywords: subgingival microbiota; chronic periodontitis; dysbiosis; deep sequencing; gingival crevicular fluid
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis; Dysbiosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — subgingival plaque sample and gingival fluid sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low severity: patient with periodontitis stage I and II
  Interventions: Other: subgingival plaque sample; Other: CGF sample
- high severity: patient with periodontitis stage III and IV
  Interventions: Other: subgingival plaque sample; Other: CGF sample

INTERVENTIONS:
Other: subgingival plaque sample — for subgingival plaque sample, on three affected sites (PD>3mm) and three healthy sites (PD≤3mm), after supra-gingival plaque removal, sterile endodontic paper points were inserted in selects pockets for 30s to collect the subgingival plaque. The material was transferred into eppendorf tube, one for affected samples and one for healthy samples.
Other: CGF sample — each site was sampled with a PerioPaper Strip® (Oraflow), and the volumes collected were measured with a Periotron® (Oraflow). Then samples of affected sites were stowed in an eppendorf tube with 120µL of PBS Tween. The same procedure was performed for the healthy sites

SUMMARY:
A new classification of periodontal diseases was created in 2018. the investigators want to know if this clinical classification is based, or not, on a biological reality. To do this, the investigators will collect data from the clinical examination (clinical assessment and radiological assessment) as well as non-invasive samples of subgingival plaque and crevicular gingival fluid (CGF). The subgingival plaque samples will be analyzed to define the microbiotic profiles of the patients and the CGF determined to define their inflammatory expression profiles. These results will then be linked to the diagnosis of severity of periodontitis.

DETAILED DESCRIPTION:
In the new classification of periodontal disease, the investigators will seek to know whether there is a specific bacterial signature associated with the severity of damage on the one hand, and the other hand, the investigators will search for cytokinic biomarkers which can be correlated with the severity of the damage.

In this study, the investigators propose to include 25 patients with periodontitis stage I and II versus stage III and IV according to Chicago classification (2018)

ELIGIBILITY:
Inclusion Criteria:

* Men and women speaking and understanding French
* Aged over 18
* with generalized periodontitis (more than 30% of affected sites)
* Requiring non-surgical periodontal therapy
* with a minimum of 12 teeth (3 per quadrant), fitted or not
* Having given his oral consent to participate in the study
* Having given his written consent to participate in a biocollection

Exclusion Criteria:

* Less than 12 teeth present (3 teeth per quadrant)
* Presence of acute oral lesions (periodontal abscesses, endodontic abscesses, infectious or mycotic lesions…)
* Presence of ulcerative-necrotic gingivitis or periodontitis
* Presence of endo-periodontal lesions
* Chronic or systemic pathology or treatment that can influence the periodontal microbiota : immunotherapy, corticosteroid therapy, biotherapy, unbalanced diabetes, acute inflammatory rheumatism, neurological impairment…
* Antibiotic during the 3 month preceding inclusion
* Psychological or linguistic disability preventing good understanding of the study
* Minors
* Major patients under legal protection
* Patients deprived of their liberty
* Pregnant or lactating woman
* Patient not affiliated to a health insurance scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient coming in consultation for generalized periodontitis .
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Microbiota analysis of subgingival plaque | through study completion, an average of 1 year
  sample analysis by microbiome sequencing with 16S technics of subgingival plaque of affected sites and healthy sites

SECONDARY OUTCOMES:
Cytokinic concentrations in CGF | through study completion, an average of 1 year
  cytokinic concentration analysis (IL1β, IL , TNFα, IL2, IL4, IL10, IL17α) in CGF of affected sites and healthy sites

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes Universitary Hospital, Nantes, Loire Atlantique, France